CLINICAL TRIAL: NCT06614829
Title: Patient Reported Experiences and Outcomes Associated with C-Section Wound Closure Bundle
Brief Title: Patient Reported Experiences and Outcomes Associated with Standard C-Section Wound Closure Versus STRATAFIX/DERMABOND PRINEO Wound Closure (CS-PREO)
Acronym: CS-PREO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: North York General Hospital (Other)
Collaborators: Johnson & Johnson (Industry)
Responsible Party: Principal Investigator, Patricia Trbovich, Badeau Family Research Chair in Patient Safety and Quality Improvement, North York General Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 0434
Record Dates: First submitted 2024-09-24; First posted 2024-09-26 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Cesarean Section; Complications, Wound, Infection (Following Delivery)
MeSH Terms: conditions — Wounds and Injuries; Infections

STUDY DESIGN:
Intervention Model Description: Parallel between group study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Control (No Intervention): This group would be receiving the standard of care.
- Bundled C-section Wound Closure (Active Comparator): Surgeons in this arm will complete elective C-section wound closure with Stratafix Sutures and the Dermabond PRINEO wound dressing.
  Interventions: Device: Stratafix Suture; Device: DERMABOND PRINEO

INTERVENTIONS:
Device: Stratafix Suture — Stratafix sutures are barbed and have an antimicrobial coating. The barbs maintain tension during and allows for knotless suturing. The antimicrobial coating inhibits bacterial colonization of the wound.
  Arms: Bundled C-section Wound Closure
Device: DERMABOND PRINEO — DERMABOND™ PRINEO™ Skin Closure System is a sterile, liquid topical skin adhesive. It also incorporates a self-adhering mesh that is applied to the approximated skin edges to provide temporary skin edge alignment until the liquid adhesive is applied to achieve skin closure. It forms a strong, flexible, waterproof microbial barrier-as long as the adhesive film remains intact-that falls off naturally after 7-14 days.
  Dermabond Prineo system will be applied to the skin for skin closure.
  Arms: Bundled C-section Wound Closure

SUMMARY:
The aim of the study is to compare outcomes between patients receiving standard C-section wound closure compared to a wound closure bundle that includes Stratafix sutures and Dermabond PRINEO.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate patient experience and patient reported outcomes following cesarean delivery in women receiving either standard wound closure or a wound closure bundle which includes both Stratfix sutures and Dermabond Prineo.

Patients in both study arms will complete established questionnaires capturing patient-reported experience measures (PREMS) and patient-reported outcome measures (PROMS).

ELIGIBILITY:
Inclusion Criteria:

1. Patient must be 18 years of age or older at time of recruitment
2. Patients opting for a planned (elective) C-Section (13-36 weeks gestation) will be eligible to consent.
3. Patients must have internet access and/or a smartphone in order to access the digital platform to complete the study questionnaires
4. Patients must speak and write in English as study questionnaires will only be provided in English
5. Patients must have coverage from the Ontario Health Insurance Plan (OHIP)

Exclusion Criteria:

1. Patients assessed by the participating surgeon with any conditions that may compromise their:

   * Ability to consent or use the virtual care platform (e.g., patients with intellectual disabilities)
   * Expectation of significant maternal complications that may affect the surgery
2. Patients who enroll in the study but have an unplanned emergency C-section

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2024-10-22 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Canadian Patient Experiences Survey - Inpatient Care + maternity questions | Assessed roughly 48-72 hours after C-section delivery
  Validated patient reported experience measure (PREM) assessing 1) communication with nurses, 2) communication with doctors, 3) involvement in decision-making and treatment options, 4) information and understanding when leaving the hospital, and 5) overall hospital experience
SCAR-Q Scores | Assessed at approximately 6 week follow-up appointment
  Validated patient reported outcome measure (PROM) assessing three domains: 1) Scar appearance, 2) Scar Symptoms, and 3) Psychosocial Impact
Diagnosed surgical site infection [Surgical site infection questionnaire completed at follow-up appointment] | Assessed at approximately 6 week follow-up appointment
  Categories include: no, superficial, deep, organ/space
Readmission to any hospital following birth [Surgical site infection questionnaire completed at follow-up appointment] | Assessed at approximately 6 week follow-up appointment
  Self-reported by patient
Antibiotic prescription for treatment of infection [Surgical site infection questionnaire completed at follow-up appointment] | Assessed at approximately 6 week follow-up appointment
  Self-reported by patient

CONTACTS AND LOCATIONS:
Locations (1):
- North York General Hospital, North York, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
Only aggregate data will be shared comparing study arms.